CLINICAL TRIAL: NCT06500767
Title: Psycho-emotional Impact of Preoperative Counselling in Cervico-carcinoma Screening
Brief Title: Psycho-emotional Impact of Preoperative Counselling in Cervico-carcinoma Screening Programs
Status: Recruiting | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: University of Torino
Record Dates: First submitted 2023-06-16; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Physiological Stress; HPV Infection; Papilloma Viral Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- counselling A: receiving counselling prior to surgery in person
- counselling B: receiving counselling prior to surgery via telephone and with a video

SUMMARY:
The communication of an altered Pap smear or positive HPV test has a strong impact on patients on a psychological level. HPV positive women are more likely to have higher level of stress, anxiety, depression and impaired sexual life.

The examiner want to establish this impact through different surveys (DASS-21 (Depression Anxiety Stress Scales); PCL-5 (Posttraumatic Stress Disorder Checklist); DTS (Dyadic Trust Scale), CDDQ (Cervical Dysplasia Distress Questionnaire) and MPI (Match Patient Inventory) from the moment the patient receives the news until after completing treatment for her intraepithelial neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* patients accessing our Colposcopy service from Prevenzione Serena program with an altered pap smear or a two-times positive HPV test
* patients with biopsy result of HSIL
* ability to fill in surveys via e-mail

Exclusion Criteria:

* previous access in our Colposcopy service
* patients not enrolled in Prevenzione Serena
* pregnant patients
* inability to fill in surveys via email
* partial or total language barrier
* denied consent to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All the patients accessing our Colposcopy service from Prevenzione Serena program with an altered pap smear or a two-times positive HPV test
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
DASS-21 (Depression Anxiety Stress Scales). | 3 to 6 months
  0 Did not apply at all 1 Applied to some degree 2 Applied to a considerable degree 3 Applied very much. I found it hard to wind down; I was aware of dryness of my mouth;I couldn't seem to experience any positive feeling at all I experienced breathing difficulty ; I found it difficult to work up the initiative to do things ;I tended to over-react to situations;I experienced trembling ;I felt that I was using a lot of nervous energy; I was worried about situations in which I might panic; I felt that I had nothing to look forward to; I found myself getting agitated; I found it difficult to relax ; I felt down-hearted and blue ; I was intolerant of anything that kept me from getting on with what I was doing ; I felt I was close to panic ; I was unable to become enthusiastic about anything ; I felt I wasn't worth much as a person ; I felt that I was rather touchy; I was aware of my heart in the absence of physical exertion ; I felt scared without reason; i felt that life was meaningless
PCL-5 (Posttraumatic Stress Disorder Checklist); | 3 to 6 months
  Not at all 0 A little bit 1 Moderately 2 Quite a bit 3 Extremely 4 Disturbing, unwanted memories of the stressful experience? Repeated dreams of it? Feeling or acting as if it were re-happening? Feeling very upset when reminded of it? Strong physical reactions when reminded? Avoiding memories or thoughts related to the experience? Avoiding external reminders? Trouble remembering important parts of it? Strong negative beliefs about yourself, others, or the world? Blaming yourself or others for the experience or its aftermath? Strong negative feelings like fear, horror, anger, guilt, or shame? Loss of interest in activities you used to enjoy? Feeling distant or cut off from others? Trouble experiencing positive feelings? Irritable behavior, angry outbursts, or acting aggressively? Taking too many risks or doing things that could harm you? Being "superalert"? Feeling easily startled? Difficulty concentrating? Trouble falling asleep?
DTS (Dyadic Trust Scale) | 3 to 6 months
  Strongly Disagree Disagree Neutral Agree Strongly Agree
  1 2 3 4 5
  Please rate the extent to which you agree or disagree with each statement:
  My partner is primarily interested in his/her own welfare. 1 2 3 4 5 There are times when my partner cannot be trusted. 1 2 3 4 5 My partner is perfectly honest and truthful with me. 1 2 3 4 5 I feel that I can trust my partner completely. 1 2 3 4 5 My partner is truly sincere in his/her promises. 1 2 3 4 5 I feel that my partner does not show me enough consideration. 1 2 3 4 5 My partner treats me fairly and justly. 1 2 3 4 5 I feel that my partner can be counted on to help me. 1 2 3 4 5 My partner behaves in a very consistent manner. 1 2 3 4 5 My partner is always honest with me.
  1 2 3 4 5
  Scoring:
  To determine the trust level, reverse score the negatively worded items (1, 2, and 6). For these items, change the scoring as follows: 1 becomes 5, 2 becomes 4, 3 stays the same, 4 becomes 2, and 5 becomes 1.
CDDQ (Cervical Dysplasia Distress Questionnaire) | 3 to 6 months
  Not at all A little bit Moderately Quite a bit Extremely 0 1 2 3 4
  Please rate how much you have been distressed by each of the following in the past week, including today:
  Worrying about the possibility of developing cancer. 0 1 2 3 4 Feeling anxious about future medical procedures. 0 1 2 3 4 Feeling down or depressed about your diagnosis. 0 1 2 3 4 Concerns about the impact of the diagnosis on your sexual relationships. 0 1 2 3 4 Feeling stressed about having to undergo regular follow-up tests. 0 1 2 3 4 Worrying about how others might react to your diagnosis. 0 1 2 3 4 Feeling upset about the uncertainty of your health status. 0 1 2 3 4 Concerns about fertility or future pregnancies. 0 1 2 3 4 Feeling isolated or alone in dealing with your diagnosis. 0 1 2 3 4 Experiencing intrusive thoughts about your condition. 0 1 2 3 4
MPI (Match Patient Inventory) | 3 to 6 months
  Strongly Disagree 1Disagree2Neutral3Agree 4Strongly Agree5Impossible to Evaluate6
  The doctor:
  Greeted me in a way that made me feel comfortable. Discussed the reason(s) that brought me here today.
  Encouraged me to express my thoughts about my health problem. Listened carefully to what I had to say.
  Understood what I had to say. the doctor explained what was done and why. Explained the necessary lab tests Discussed treatment options with me. Gave me all the information I wanted.Checked whether the treatment plan(s) were acceptable to me. Gave explanations regarding any medications, including possible side effects.
  Encouraged me to ask questions. Answered my questions and concerns. Involved me in decisions as much as I wanted. Discussed the next steps, including any follow-up plans. Made sure I understood everything.
  Showed interest and concern for me as a person. Spent the right amount of time with me. Overall, I am satisfied with today's visit with the doctor

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Sant'Anna, Turin, TO, Italy